CLINICAL TRIAL: NCT05310123
Title: Investigation of AC-11® Supplementation in Reversing Epigenetic Markers of Biological Aging Including Those Related to Telomere Length
Brief Title: AC-11 Supplement and Biological Aging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TruDiagnostic (Industry)
Collaborators: Optigenex, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OI-AC11-001
Record Dates: First submitted 2022-03-02; First posted 2022-04-04 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: prospective, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AC-11 (Experimental): 6 months of treatment with AC-11
  Interventions: Dietary Supplement: AC-11

INTERVENTIONS:
Dietary Supplement: AC-11 — 6-months of treatment with AC-11

SUMMARY:
This is a prospective non-randomized clinical study of 24 patients to evaluate the effects of the AC-11®. The study will evaluate the effectiveness of the supplement's ability to reverse epigenetic markers of biological age. The duration of the study will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of any ethnicity.
2. Age Range 55 years and older
3. The patient must be able to comply with the treatment plan and laboratory tests

Exclusion Criteria:

1. Neoplastic cancer within 5 years prior to screening, except for cutaneous basal cell or squamous cell cancer resolved by excision
2. No immune system issues or immunodeficiency disease
3. No history of viral illness which could be reactivated by immune downregulation
4. Presence of clinically significant acute or unstable cardiovascular and cerebrovascular (stroke)
5. Diagnosis of a transient ischemic attack in the 6 months prior to screening
6. Patients infected with hepatitis C or HIV
7. Patients with Body Mass Index (BMI) > 40 kg/m2
8. Presence of active infection
9. Any other illness, psychiatric disorder, alcohol or chemical dependence that in the opinion of the investigator would render a patient unsuitable to participate in the study
10. Unable or unwilling to provide a required blood sample for testing
11. As for the male-participants they are recommended to avoid fertilization for the first 6 months after the clinical trial.
12. If the patient has previously used AM/PM HealthSpan system supplements at any time before the start of the trial.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Methylation age clock testing | Change in epigenetic age from baseline to 6 months
  Epigenetic testing
Telomere Test | Change in telomere length from baseline to 6 months
  Epigenetic testing

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Gallegos, Principal Investigator — Thrive Medicine Clinic
Locations (1):
- Thrive Medicine Clinic, Sugar Land, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guthrie OW, Xu H. Reduced Phosphorylation of Histone Variant H2Ax in the Organ Of Corti Is Associated With Otoprotection from Noise Injury. Otolaryngology 2013; 3:131.